CLINICAL TRIAL: NCT05504759
Title: Evaluation of the Efficacy of Dry Needling Treatment of Wrist Extensor Muscles in the Treatment of Lateral Epicondylitis
Brief Title: Efficacy of Dry Needling in the Treatment of Lateral Epicondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Emre Ata, Assoc Prof, Associate Proffesor, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2166
Record Dates: First submitted 2022-03-31; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Lateral Epicondylitis
Keywords: tennis elbow; dry needling
MeSH Terms: conditions — Tennis Elbow | interventions — Splints; Steroids; Dry Needling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): 2 weeks rest protocol + standardized exercise program
  Interventions: Other: splint
- Group 2 (Experimental): local steroid injection + 2 weeks rest protocol + standardized exercise program
  Interventions: Other: splint; Other: steroid
- Group 3 (Experimental): dry needling of forearm extensor muscles + 2 weeks rest protocol + standardized exercise program
  Interventions: Other: splint; Other: dry needling

INTERVENTIONS:
Other: splint — Resting is the first step of treatment in lateral epicondylitis. Patients will be given a 2 weeks rest protocol (works that may cause strain on the wrist and increase elbow pain will be described and it will be advised to stay away, and a home exercise program will be prepared, which includes the use of a resting splint during the daytime for 2 weeks). The goal of exercise therapy will be to stretch the muscles, strengthen them and maintain flexibility. Home exercises during the treatment of lateral epicondylitis will be beneficial when performed twice a day for at least three months, and stretching exercises will be performed first, and then strengthening exercises will be started in a controlled manner.
Other: steroid — Betamethasone Dipropionate + Betamethasone Sodium Phosphate-1 ml will be administered once at the beginning of the study to patients who will receive steroid injection, one of the local injection treatments. Steroid injection will be applied to the most sensitive point on the lateral epicondyle. Afterwards, patients will be given a 2 weeks rest protocol (works that may cause strain on the wrist and increase elbow pain will be described and it will be advised to stay away, and a home exercise program will be prepared, which includes the use of a resting splint during daytime hours for 2 weeks). The goal of exercise therapy will be to stretch the muscles, strengthen them and maintain flexibility. Home exercises during the treatment of lateral epicondylitis will be beneficial when performed twice a day for at least three months, and stretching exercises will be performed first, and then strengthening exercises will be started in a controlled manner.
  Arms: Group 2
Other: dry needling — The needle will be guided to painful trigger points detected by palpation. Stainless steel 25x30 mm needles will be used for dry needling. Dry needle treatment will be applied to the painful trigger points in the forearm extensor group muscles with the stick-pull technique, 1 session per week, for a total of 2 sessions. Afterwards, the patients will be given a 2 weeks rest protocol (works that may strain the wrist and increase elbow pain will be described and it will be advised to stay away, and a home exercise program will be prepared, which includes the use of a resting splint during the daytime for 2 weeks). The purpose of exercise therapy will be to stretch the muscles, strengthen them and maintain flexibility. During the treatment of lateral epicondylitis, home exercises will be beneficial when performed twice a day for at least three months, and stretching exercises will be performed first, and then strengthening exercises will be started in a controlled manner.
  Arms: Group 3

SUMMARY:
In this study, investigators aimed to investigate the effects of rest, steroid injection and dry needling treatments, which are frequently used in the treatment of patients diagnosed with lateral epicondylitis (tennis elbow), on the pain and functional status of the patients.

DETAILED DESCRIPTION:
Lateral epicondylitis is one of the most common painful conditions of the arm, characterized by pain in the lateral epicondyle where the wrist extensors muscles originate and on the extensor muscle surface of the forearm, and is also called tennis elbow. The incidence of lateral epicondylitis has been reported as 1-3%. The age of onset is between 35 and 50, and it is more common in men. Mostly the dominant arm is affected, rarely bilateral. It may occur as a result of repetitive and difficult wrist extension. Tenderness in the lateral epicondyle, pain that can be revealed with resistant wrist extension and middle finger extension, decrease in grip strength and significant limitation in daily living activities are the main findings. The repetition of the movement is more important than the force required to perform the movement in the development of the symptoms. Extensor muscles are under extreme stress in those who work in jobs that require continuous rotation of the wrist, such as grasping, supination, and pronation, or in these types of sports. As a result of forcing, soft tissues such as muscles, ligaments and tendons in the forearm cannot meet the load they are exposed to, and thus symptoms occur. Although it originates from the muscle extensor carpi radialis brevis (ECRB), where pathological changes are primarily seen; It can also be seen at the origin of the extensor carpi radialis longus (ECRL) and extensor digitorum communis (EDK) muscles. Myofascial trigger points formed in the forearm extensor group muscles are frequently detected during examination.

The basic principles of treatment in lateral epicondylitis are to relieve pain, accelerate the healing process, reduce overloads on the arm, and enable the patient to return to daily life activities. Conservative treatment options are rest, splint, ice application, electrotherapy, massage, manipulation, mobilization, exercise and medical therapy.

When investigators examine the literature, although there are many studies on conservative methods and steroid injection in the treatment of lateral epicondylitis; investigatorsfound several studies on the effectiveness of dry needling in lateral epicondylitis. In the current study, the efficacy of dry needling was compared with the conservative method, which is only the first-line treatment. In addition, in these studies, dry needling was applied to the musculeutendinous junction. Investigators observed that lateral epicondylitis is a disease that is activated by tendinopathy and can cause multiple painful tender points and tight bands in the forearm muscles. In this context, investigators think that more studies are needed on the effectiveness of dry needling in lateral epicondylitis. In this study, investigators aimed to investigate the effects of rest, steroid injection and dry needling treatments, which are frequently used in the treatment of patients diagnosed with lateral epicondylitis (tennis elbow), on the pain and functional status of the patients.

The first stage of treatment is rest, orthoses can also be used in this regard. The use of a forearm support band and a splint to keep the wrist at 20 degrees of extension also helps to keep the extensor muscles in a relaxed position, resting these muscles.

At the end of the 2-week rest period, patients are given strengthening and stretching exercises. Strengthening the wrist extensors increases the tolerance of the damaged attachment to repetitive and resistant movement. Mills maneuver, that is, extension of the elbow, pronation of the forearm, flexion of the wrist and ulnar deviation as a stretching exercise for 30-45 seconds. applicable. The goal with stretching is to lengthen the scar tissue.

Ultrasound, iontophoresis, laser, interference currents, electrical stimulation, ESWT are physical therapy methods used in lateral epicondylitis. In addition to the analgesic effects of these treatment methods, their contribution to the healing process of the damaged tissue has also been reported.In addition, various injection methods (steroid injection, prolotherapy, platelet rich plasma (PRP), dry needling) are also used in the routine treatment of lateral epicondylitis.

Many treatment methods have been reported in the studies on the treatment of lateral epicondylitis, but in general, insufficient number of patients and short follow-up periods are stated as the missing aspects of the studies. The aim of our study is to evaluate in detail the methods used in the routine for treatment, which do not have side effects and are comfortable, and compare the superiority of the methods to each other. In addition, by examining the efficacy of treatment with sufficient number of patients and follow-up period in our study; It is aimed to contribute to the literature by evaluating the methods in terms of safety, effectiveness, efficiency, accessibility, quality and determining the most appropriate methods for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-65 years with pain in the lateral humeral epicondyle region for at least 6 weeks
2. Patients with pain on palpation of the lateral humeral epicondyle and patients with lateral epicondyle pain manifested by at least one of the provocative tests, such as resistant middle finger extension or resistant wrist extension or passively stretching the wrist extensors
3. Patients with painful trigger points detected by palpation in the extensor group muscles of the forearm

Exclusion Criteria:

1. History of upper extremity trauma or surgery
2. History of arthritis in the upper extremity
3. Patients with EMG-proven entrapment neuropathy in the upper extremity
4. Patients with cervical radiculopathy
5. History of interventional procedures such as physical therapy or steroid injection for lateral epicondylitis in the last 3 months
6. Pregnancy and pregnancy
7. Patients with complaint duration less than 6 weeks
8. Having mental (intelligence-related) problems, limitation of cooperation-orientation (being aware of time and space and having communication skills)
9. <18 years, >65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-06-02 (Estimated); Study Completion 2023-08-02 (Estimated)

PRIMARY OUTCOMES:
change in elbow pain after treatment as assessed by vas | before treatment, second-month control after treatment
  Elbow pain will be measured with the Visual Analog Scale (VAS).The Visual Analog Scale (VAS) is used to convert some values that cannot be measured numerically. Two end definitions of the parameter to be evaluated are written at the two ends of a 100 mm line, and the patient is asked to indicate where on this line their situation is appropriate by drawing a line or by placing a dot or pointing. For example, for pain, I have no pain at one end and very severe pain at the other end and the patient marks his/her current state on this line. The length of the distance from the point where there is no pain to the point marked by the patient indicates the patient's pain.

SECONDARY OUTCOMES:
Hand grip strength | before treatment, second-month control after treatment.
  It will be evaluated with the Jamar hydraulic hand dynamometer.The purpose of this test is to test the maximum isometric contraction strength of the hand and forearm muscles. A hand grip dynamometer is required to perform the test (such as Jamar™, Camry™, Smedley™). Dynamometer Examples Grip strength should be evaluated while the patient is sitting in the chair. The elbows are kept close to the body and at 90° flexion. The wrist is in neutral. The person to be measured is asked to grasp the dynamometer and squeeze it as hard as he can. The test result is determined by calculating the average of the three measurements. Norm values for measurement: 47-40kg for men aged 20-69 (left hand 2 kg less) 30-24kg for women (1.5-2kg less for left hand)

CONTACTS AND LOCATIONS:
Overall Officials: Emre Ata, Ass.Prof., Principal Investigator — Sultan II. Abdulhamidhan Training and Research Hospital
Locations (1):
- Sultan 2. Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Türkiye)